CLINICAL TRIAL: NCT03897816
Title: Maternal Mood, Anxiety or Personality Disorders and Their Offspring Mental Outcomes
Brief Title: Maternal Psychopathology and Offspring Mental Health (PSI_PER)
Acronym: PSI_PER
Status: Completed | Type: Observational
Sponsor: University of Milano Bicocca (Other)
Responsible Party: Sponsor
Other Study IDs: 981
Record Dates: First submitted 2019-03-29; First posted 2019-04-01 (Actual); Last update posted 2019-04-04 (Actual); Status verified 2019-04

CONDITIONS: Intergenerational Relations
Keywords: personality disorders; anxiety disorders; mood disorders
MeSH Terms: conditions — Personality Disorders; Anxiety Disorders; Mood Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- "PERINATAL": Pregnant women consecutively referred and admitted to the Perinatal Psychiatric Outpatient Department
- "OUTPTS": Pregnant women belonging to the Outpatients Psychiatric Department who did not have psychiatric issues linked to their pregnancy or in the relationship with their children
- Healthy controls: Pregnant women the general population, with no history of mental health issues

SUMMARY:
Pregnant women consecutively referred to the Perinatal Psychiatric Outpatient Department, those in charge of the Psychiatric Outpatient Department and pregnant healthy controls from the general population will be recruited on a voluntary basis. Mothers will be tested with the EPDS, BAI, BDI, WHOQOL, SCID II and CTQ; their children will be tested with the CBCL between 18 months and 5 years.

DETAILED DESCRIPTION:
in order to attest possible psychic outcomes in offspring of mothers affected by psychiatric disorders due to maternal psychopathology (with an in-depth evaluation about the role of maternal personality disorders), the investigators recruit all the women consecutively referred and admitted to the Perinatal Psychiatric Outpatient Department from January, 2011 to December, 2016, due to the manifestation of psychic suffering during pregnancy.

During their first appointment, patients are routinely administered the Structured Clinical Interview for DSM-IV Axis II Disorders (SCID II), Childhood Trauma Questionnaire (CTQ), World Health Organization Quality of Life Instruments (WHOQOL-BREF), Edinburgh Postnatal Depression Scale (EPDS), Beck Depression Interview (BDI) and Beck Anxiety Interview (BAI). The Mini-International Neuropsychiatric Interview (M.I.N.I.) is used to confirm clinical diagnosis.

As a control samples, the investigators recruited pregnant patients belonging to the Outpatients Psychiatric Department who did not have psychiatric issues linked to their pregnancy or in the relationship with their children and pregnant healthy controls among the general population, with no history of mental health issues. Controls were tested as the clinical sample.

All the patients will be asked to complete a caregiver report form, the Child Behavior Checklist (CBCL), once their children were at least 18 months old.

ELIGIBILITY:
Inclusion Criteria:

pregnancy; adequate comprehension; acceptance on a voluntary basis.

Exclusion Criteria:

incapacity; acute psychosis.

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — pregnant women
Study Population: the population is composed by women referred to the Perinatal Psychiatric Outpatient Department, those in charge of the Psychiatric Outpatient Department and pregnant healthy controls from the general population.
Sampling Method: Non-Probability Sample
Enrollment: 450 (Actual)
Dates: Start 2011-01-01 (Actual); Primary Completion 2016-03-15 (Actual); Study Completion 2019-02-01 (Actual)

PRIMARY OUTCOMES:
offspring mental outcomes | 18 months-5 years old
  Mothers are given the Child Behavior Checklist (CBCL), a widely used caregiver report form identifying problem behavior in children. For the preschool version of the CBCL (CBCL/1½-5), parents or others who interact with the child in regular contexts rate the child's behavior. Respondents rate the child's behavior on a 3-point scale (not true, somewhat or sometimes true, and very true or often true), and are instructed to rate the behavior as it occurs now or within the previous two months. This delineation differs from the instructions on other age-versions, due to the fact that rapid development and behavioral changes in the preschool age range are common. The preschool checklist contains 100 questions about behavior problems.
  CBCL scores are divided in: "emotionally reactive", "anxious/depressed", "somatic complaints", "withdrawn", "sleep problems", "attention problems", "aggressive behavior", "externalize", "internalize", "other problems", "total".

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Bloch M, Schmidt PJ, Danaceau M, Murphy J, Nieman L, Rubinow DR. Effects of gonadal steroids in women with a history of postpartum depression. Am J Psychiatry. 2000 Jun;157(6):924-30. doi: 10.1176/appi.ajp.157.6.924. PMID 10831472
- [Background] Mehta D, Newport DJ, Frishman G, Kraus L, Rex-Haffner M, Ritchie JC, Lori A, Knight BT, Stagnaro E, Ruepp A, Stowe ZN, Binder EB. Early predictive biomarkers for postpartum depression point to a role for estrogen receptor signaling. Psychol Med. 2014 Aug;44(11):2309-22. doi: 10.1017/S0033291713003231. Epub 2014 Feb 5. PMID 24495551
- [Background] Couto TC, Brancaglion MY, Alvim-Soares A, Moreira L, Garcia FD, Nicolato R, Aguiar RA, Leite HV, Correa H. Postpartum depression: A systematic review of the genetics involved. World J Psychiatry. 2015 Mar 22;5(1):103-11. doi: 10.5498/wjp.v5.i1.103. PMID 25815259
- [Background] Guintivano J, Arad M, Gould TD, Payne JL, Kaminsky ZA. Antenatal prediction of postpartum depression with blood DNA methylation biomarkers. Mol Psychiatry. 2014 May;19(5):560-7. doi: 10.1038/mp.2013.62. Epub 2013 May 21. PMID 23689534
- [Background] Ruiz SK, Harris SJ, Martinez P, Gold PM, Klimes-Dougan B. Young adult's attachment style as a partial mediator between maternal functioning and young adult offsprings' functioning. J Affect Disord. 2018 May;232:393-399. doi: 10.1016/j.jad.2017.12.034. Epub 2018 Jan 9. PMID 29522959
- [Background] Stein A, Pearson RM, Goodman SH, Rapa E, Rahman A, McCallum M, Howard LM, Pariante CM. Effects of perinatal mental disorders on the fetus and child. Lancet. 2014 Nov 15;384(9956):1800-19. doi: 10.1016/S0140-6736(14)61277-0. Epub 2014 Nov 14. PMID 25455250
- [Background] Matijasevich A, Murray J, Cooper PJ, Anselmi L, Barros AJ, Barros FC, Santos IS. Trajectories of maternal depression and offspring psychopathology at 6 years: 2004 Pelotas cohort study. J Affect Disord. 2015 Mar 15;174:424-31. doi: 10.1016/j.jad.2014.12.012. Epub 2014 Dec 13. PMID 25553403
- [Background] Sellers R, Collishaw S, Rice F, Thapar AK, Potter R, Mars B, Harold GT, Smith DJ, Owen MJ, Craddock N, Thapar A. Risk of psychopathology in adolescent offspring of mothers with psychopathology and recurrent depression. Br J Psychiatry. 2013 Feb;202:108-14. doi: 10.1192/bjp.bp.111.104984. Epub 2012 Oct 11. PMID 23060622
- [Background] Wisner KL, Sit DK, McShea MC, Rizzo DM, Zoretich RA, Hughes CL, Eng HF, Luther JF, Wisniewski SR, Costantino ML, Confer AL, Moses-Kolko EL, Famy CS, Hanusa BH. Onset timing, thoughts of self-harm, and diagnoses in postpartum women with screen-positive depression findings. JAMA Psychiatry. 2013 May;70(5):490-8. doi: 10.1001/jamapsychiatry.2013.87. PMID 23487258
- [Background] Challacombe F, Salkovskis P. A preliminary investigation of the impact of maternal obsessive-compulsive disorder and panic disorder on parenting and children. J Anxiety Disord. 2009 Oct;23(7):848-57. doi: 10.1016/j.janxdis.2009.04.002. Epub 2009 Apr 23. PMID 19464141
- [Background] Low NC, Dugas E, Constantin E, Karp I, Rodriguez D, O'Loughlin J. The association between parental history of diagnosed mood/anxiety disorders and psychiatric symptoms and disorders in young adult offspring. BMC Psychiatry. 2012 Nov 5;12:188. doi: 10.1186/1471-244X-12-188. PMID 23126640
- [Background] Martini J, Knappe S, Beesdo-Baum K, Lieb R, Wittchen HU. Anxiety disorders before birth and self-perceived distress during pregnancy: associations with maternal depression and obstetric, neonatal and early childhood outcomes. Early Hum Dev. 2010 May;86(5):305-10. doi: 10.1016/j.earlhumdev.2010.04.004. Epub 2010 May 23. PMID 20547016
- [Background] Black DW, Gaffney GR, Schlosser S, Gabel J. Children of parents with obsessive-compulsive disorder -- a 2-year follow-up study. Acta Psychiatr Scand. 2003 Apr;107(4):305-13. doi: 10.1034/j.1600-0447.2003.02182.x. PMID 12662254
- [Background] Castelli RD, Quevedo Lde A, Coelho FM, Lopez MA, da Silva RA, Bohm DM, Souza LD, de Matos MB, Pinheiro KA, Pinheiro RT. Cognitive and language performance in children is associated with maternal social anxiety disorder: A study of young mothers in southern Brazil. Early Hum Dev. 2015 Dec;91(12):707-11. doi: 10.1016/j.earlhumdev.2015.10.002. Epub 2015 Nov 16. PMID 26544906
- [Background] Gaynes BN, Gavin N, Meltzer-Brody S, Lohr KN, Swinson T, Gartlehner G, Brody S, Miller WC. Perinatal depression: prevalence, screening accuracy, and screening outcomes. Evid Rep Technol Assess (Summ). 2005 Feb;(119):1-8. doi: 10.1037/e439372005-001. No abstract available. PMID 15760246
- [Background] Munk-Olsen T, Laursen TM, Pedersen CB, Mors O, Mortensen PB. New parents and mental disorders: a population-based register study. JAMA. 2006 Dec 6;296(21):2582-9. doi: 10.1001/jama.296.21.2582. PMID 17148723
- [Background] Paulson JF, Bazemore SD. Prenatal and postpartum depression in fathers and its association with maternal depression: a meta-analysis. JAMA. 2010 May 19;303(19):1961-9. doi: 10.1001/jama.2010.605. PMID 20483973
- [Background] Lindahl V, Pearson JL, Colpe L. Prevalence of suicidality during pregnancy and the postpartum. Arch Womens Ment Health. 2005 Jun;8(2):77-87. doi: 10.1007/s00737-005-0080-1. Epub 2005 May 11. PMID 15883651
- [Background] Earls MF; Committee on Psychosocial Aspects of Child and Family Health American Academy of Pediatrics. Incorporating recognition and management of perinatal and postpartum depression into pediatric practice. Pediatrics. 2010 Nov;126(5):1032-9. doi: 10.1542/peds.2010-2348. Epub 2010 Oct 25. PMID 20974776
- [Background] Bosanquet K, Bailey D, Gilbody S, Harden M, Manea L, Nutbrown S, McMillan D. Diagnostic accuracy of the Whooley questions for the identification of depression: a diagnostic meta-analysis. BMJ Open. 2015 Dec 9;5(12):e008913. doi: 10.1136/bmjopen-2015-008913. PMID 26656018
- [Background] Wisner KL, Parry BL, Piontek CM. Clinical practice. Postpartum depression. N Engl J Med. 2002 Jul 18;347(3):194-9. doi: 10.1056/NEJMcp011542. No abstract available. PMID 12124409
- [Background] Goodman JH. Postpartum depression beyond the early postpartum period. J Obstet Gynecol Neonatal Nurs. 2004 Jul-Aug;33(4):410-20. doi: 10.1177/0884217504266915. PMID 15346666
- [Background] Byatt N, Levin LL, Ziedonis D, Moore Simas TA, Allison J. Enhancing Participation in Depression Care in Outpatient Perinatal Care Settings: A Systematic Review. Obstet Gynecol. 2015 Nov;126(5):1048-1058. doi: 10.1097/AOG.0000000000001067. PMID 26444130